CLINICAL TRIAL: NCT02762279
Title: Assessment of Esophageal Pressure Reliability to Estimate Pleural Pressure in Critically Ill Children
Acronym: APPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Dr Guillaume Emeriaud, MD PHD, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUSJ 2016-1238
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Mechanical Ventilation
Keywords: Mechanical ventilation; Children; Esophageal Pressure; Pleural Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): 1. Patient baseline characteristics will be collected.
  2. Specific nasogastric tube installation: a specific nasogastric tube equipped with pressure transducers (Gaeltec® probe) will be installed.
  3. Connection of a pressure transducer to the existing chest-tube.
  4. Simultaneous recordings of PES (Gaeltec®), PPL, PAW, respiratory volume and flow (5 minutes).
  5. Removal of the Gaeltec® probe, and repositioning of the pre-existing nasogastric tube in the esophagus for PES measurement.
  6. Simultaneous recordings of PES (feeding tube), PPL, PAW, respiratory volume and flow (5 minutes).
  7. Repositioning of the nasogastric tube in the stomach, and disconnection of the different recording equipment.
  Interventions: Other: esophageal and pleural pressure measurement

INTERVENTIONS:
Other: esophageal and pleural pressure measurement — Esophageal pressure will be monitored by a dedicated catheter and pleural pressure will be measured into the chest tube already in place

SUMMARY:
Background During ventilatory assistance, optimization of settings is critical to allow a personalized support and avoid over- or under-assistance. But little data are available in clinical practice to guide the adjustment of the support. In adults, esophageal pressure (PES) has been shown to be a reliable surrogate of pleural pressure (PPL) and clinical studies suggest that PES may be useful to guide the management of mechanical ventilation. In children, the PES measurement could have similar potential benefits, but beforehand the reliability of PES to estimate PPL needs to be assessed.

Objective The primary objective of this study is to validate the reliability of PES directly monitored using a miniature catheter tip pressure transducer (Gaeltec® system) to estimate PPL, when compared to a gold standard, i.e the direct PPL measurement in situ.

Method This is a prospective single center study. Children <18 years old, hospitalized in the pediatric intensive care unit, requiring invasive ventilation and with at least one chest tube will be included.

Protocol A pressure transducer will be connected to the existing chest-tube and PES (measured by Gaeltec® and feeding tube), PPL, PAW, respiratory volume and flow will be simultaneously recorded.

Expected results We expect that the PES-based methods will provide an accurate estimation of PPL. Once this tool validated, PES could be helpful to optimize mechanical ventilation in children, and further interventional trials would be warranted to evaluate if its use could allow a reduction of the ventilation support duration.

ELIGIBILITY:
Inclusion Criteria:

* Children <18 years old, hospitalized in the pediatric intensive care unit;
* Requiring invasive ventilation for more than 4 hours according to the prescription of the attending physician;
* With at least one chest tube.

Exclusion Criteria:

* Contraindications to the placement of a new nasogastric tube (e.g. bilateral phrenic paralysis, trauma or recent surgery in cervical or nasopharyngeal regions, severe coagulation disorder);
* Hemodynamic instability, as defined by the treating team, and the absence of recent (<4 hours) increase in the flow of dopamine, epinephrine, norepinephrine, or dobutamine;
* Respiratory instability defined as a severe respiratory failure requiring FiO2 > 60%, or PaCO2 > 80 mmHg on blood gas in the last hour;
* Persistent pleural effusion or pneumothorax despite the chest-tube;
* Bronchopleural fistula;
* Recent (<12 hours) thoracic hemorrhage;
* Delayed sternal closure at the time of study;
* Significant pericardial effusion;
* Absence of parental or tutor consent;
* Patient for whom a limitation of life support treatments is discussed or decided.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
End-expiratory esophageal | Up to 2 hours from the beginning of the study
  End-expiratory PES and PL, calculated as the mean value of 10 consecutive breaths, during a stable period with no intervention or artifacts;
Pleural pressure | Up to 2 hours from the beginning of the study
  PPL, directly measured in the existing chest tubes, and calculated as the mean value of 10 consecutive breaths, during a stable period with no intervention or artifacts.
transpulmonary pressures | Up to 2 hours from the beginning of the study

SECONDARY OUTCOMES:
The Elastance-derived end-inspiratory transpulmonary pressure | Up to 2 hours from the beginning of the study
  The Elastance-derived end-inspiratory transpulmonary pressure, calculated as: PAW at end-inspiration x EL/ERS (EI and ERS being the respective elastances of the lung and the respiratory system, estimated on the esophageal and airway Pressure-Volume curves);

CONTACTS AND LOCATIONS:
Locations (1):
- St. Justine's Hospital, Montreal, Quebec, Canada